CLINICAL TRIAL: NCT02805998
Title: Research on Expecting Moms and Sleep Therapy
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-19537
Record Dates: First submitted 2016-06-07; First posted 2016-06-20 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Therapeutics

ARMS (2):
- Web-based CBT-I (Experimental): Sleepio delivers CBT-I through 6 weekly web-sessions. Treatment content is based on CBT for insomnia manuals and includes a behavioral component (sleep restriction, stimulus control, and relaxation), a cognitive component (paradoxical intention, cognitive restructuring, mindfulness, positive imagery, putting the day to rest) and an educational component (psycho-education, sleep hygiene).
  Interventions: Behavioral: Web-based CBT-I; Other: Treatment as Usual
- Treatment as Usual (Other): Our control condition was designed to reflect standard care for insomnia patients. No limits are placed on receiving non-study treatment, including medication or psychotherapy. Use of non-study treatment will be tracked.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Web-based CBT-I
  Arms: Web-based CBT-I
Other: Treatment as Usual

SUMMARY:
The overarching goal is to utilize a randomized control design to examine efficacy of web-based cognitive behavior therapy (CBT-I) plus treatment as usual compared to treatment as usual alone for insomnia and depression outcomes among pregnant women with insomnia at high risk for depressive relapse/recurrence (n=208).

DETAILED DESCRIPTION:
Depression in pregnancy ("antenatal depression") is common and associated with acute and long-lasting adverse consequences for women and offspring. Insomnia is a risk factor for depression in general populations, and poor sleep quality is linked to increased depression among antenatal women. There have been no randomized control trials investigating nonpharmacological insomnia treatment on antenatal insomnia and depression outcomes. Many pregnant women use the Internet to seek pregnancy-related information, and report a preference for mental health care within the home or obstetrics clinic. The overarching goal is to utilize a randomized control design to examine efficacy of web-based cognitive behavior therapy for insomnia and depression outcomes (CBT-I) compared to treatment as usual (TAU) among pregnant women at risk for depression (n=208). Participants will be recruited nationally to complete study questionnaires at five timepoints through pregnancy and 6 months postpartum. Participants randomized to CBT-I will receive access to 6 weekly CBT-I web-sessions and treatment as usual. Participants randomized to treatment as usual will receive usual care and will be given access to Sleepio upon study completion. Our specific aims are:

1. To evaluate feasibility and acceptability of CBT-I for pregnant women.
2. To test whether participants receiving CBT-I show improvement in sleep compared to TAU participants.
3. To examine whether participants randomized to CBT-I will experience improved depressive outcomes compared to TAU.
4. To explore the impact of CBT-I on birth outcomes.

There is strong conceptual basis to predict the potential benefit of this approach for pregnant women. Targeting risk factors for antenatal depression may have significant public health benefits.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant up to 28 weeks gestation,
2. 18 years of age or older,
3. Meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Insomnia disorder as determined by the Sleep Condition Indicator (SCI) or Insomnia Severity Index (ISI) score ≥ 11
4. regular access to a web-enabled computer, tablet, or smart phone.

Exclusion Criteria:

1. Probable major depression (Edinburgh Postnatal Depression Scale (EPDS) score ≥ 15),
2. self-reported bipolar disorder,
3. self-reported history of psychosis,
4. active suicidality defined as scoring > 1 on EPDS item 10 or report of a specific suicide plan or recent attempt,
5. shift work employee,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Felder, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Felder JN, Epel ES, Neuhaus J, Krystal AD, Prather AA. Randomized controlled trial of digital cognitive behavior therapy for prenatal insomnia symptoms: effects on postpartum insomnia and mental health. Sleep. 2022 Feb 14;45(2):zsab280. doi: 10.1093/sleep/zsab280. PMID 34850238
- [Derived] Felder JN, Epel ES, Neuhaus J, Krystal AD, Prather AA. Efficacy of Digital Cognitive Behavioral Therapy for the Treatment of Insomnia Symptoms Among Pregnant Women: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):484-492. doi: 10.1001/jamapsychiatry.2019.4491. PMID 31968068

RESULTS

PARTICIPANT FLOW:
Groups:
- Web-based CBT-I: Sleepio delivers cognitive behavior therapy for insomnia (CBT-I) through 6 weekly web-sessions. Treatment content is based on CBT for insomnia manuals and includes a behavioral component (sleep restriction, stimulus control, and relaxation), a cognitive component (paradoxical intention, cognitive restructuring, mindfulness, positive imagery, putting the day to rest) and an educational component (psycho-education, sleep hygiene).
  Web-based CBT-I
  Treatment as Usual
- Treatment as Usual: Our control condition was designed to reflect standard care for insomnia patients. No limits are placed on receiving non-study treatment, including medication or psychotherapy. Use of non-study treatment will be tracked.
  Treatment as Usual
Period: Overall Study
Arm/Group | Web-based CBT-I | Treatment as Usual
Started | 105 | 103
Completed (Completed is defined as completing the primary outcome measure at the post-intervention timepoint.) | 91 | 94
Not Completed | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Web-based CBT-I: Sleepio delivers CBT-I through 6 weekly web-sessions. Treatment content is based on CBT for insomnia manuals and includes a behavioral component (sleep restriction, stimulus control, and relaxation), a cognitive component (paradoxical intention, cognitive restructuring, mindfulness, positive imagery, putting the day to rest) and an educational component (psycho-education, sleep hygiene).
  Web-based CBT-I
  Treatment as Usual
- Total: Total of all reporting groups
Arm/Group | Web-based CBT-I | Treatment as Usual | Total
Number analyzed (Participants) | 105 | 103 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (3.38) | 33.2 (4.0) | 33.6 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 103 | 208
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic | 100 | 93 | 193
  Hispanic | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 105 | 103 | 208
Gestational age at screening [Mean (Standard Deviation); unit: weeks] | 17.1 (6.4) | 18.07 (6.3) | 17.6 (6.3)
Income greater than or equal to 100,000 dollars [Count of Participants; unit: Participants] | 71 | 70 | 141
Married or cohabitating [Count of Participants; unit: Participants] | 100 | 96 | 196
Primiparous [Count of Participants; unit: Participants] | 46 | 66 | 112
Insomnia symptom severity [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity Index (ISI). Scores on the ISI range from 0 to 28, with higher scores indicating more severe insomnia.
  units on a scale | 14.52 (3.26) | 14.19 (3.72) | 14.36 (3.49)
Percentage of sleep efficiency [Mean (Standard Deviation); unit: percentage] — Daily sleep diaries were used to measure sleep efficiency. Sleep efficiency was calculated by dividing the amount of time sleeping by the amount of time spent in bed. Sleep efficiency ranges from 0 to 100 percent, with higher scores indicating better outcomes.
  percentage | 72.22 (12.35) | 74.19 (11.96) | 73.20 (12.17)
Nightly sleep duration [Mean (Standard Deviation); unit: hours] | 6.68 (1.13) | 6.84 (1.23) | 6.76 (1.18)
Global sleep quality [Mean (Standard Deviation); unit: units on a scale] — Global sleep quality was measured using the Pittsburgh Sleep Quality Index (PSQI). Scores range from 0 to 21, with higher scores indicating worse global sleep quality.
  units on a scale | 9.52 (2.74) | 9.47 (3.02) | 9.50 (2.87)
Insomnia caseness [Count of Participants; unit: Participants] — Insomnia caseness (i.e., whether a participant met the Diagnostic and Statistical Manual for Mental Disorders, Fifth Edition criteria for insomnia disorder) was assessed by the Sleep Condition Indicator (SCI), which is an eight-item rating scale to screen for an insomnia diagnosis. Insomnia caseness was determined by a complex scoring algorithm for the SCI.
  Participants | 54 | 41 | 95
Depressive symptom severity [Mean (Standard Deviation); unit: units on a scale] — Depressive symptom severity was assessed using the Edinburgh Postnatal Depression Scale (EDPS). Scores on the EPDS range from 0 to 30, with higher scores indicating greater depressive symptom severity.
  units on a scale | 7.79 (4.05) | 7.24 (3.77) | 7.52 (3.91)
Anxiety symptom severity [Mean (Standard Deviation); unit: units on a scale] — Anxiety symptom severity was assessed using the Generalized Anxiety Disorder Scale-7. Scores range from 0 to 21, with higher scores indicating greater anxiety symptom severity.
  units on a scale | 5.43 (3.55) | 4.81 (3.23) | 5.12 (3.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index Scale Score
Description: Insomnia Severity Index (ISI). Scores on the ISI range from 0 to 28, with higher scores indicating more severe insomnia.
Time Frame: Baseline to post-intervention (10 weeks post-randomization)
Population: The number of participants analyzed is fewer than the number of participants who completed each arm of the study due to 23 participants being lost-to-follow up and not completing the ISI at post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based CBT-I | Treatment as Usual
Number analyzed (Participants) | 91 | 94
units on a scale | -6.054945 (4.347062) | -2.212766 (4.699285)

2. Secondary Outcome: Change in Percentage of Sleep Efficiency, as Determined by Daily Sleep Logs
Description: Daily sleep diaries were used to measure percentage of sleep efficiency. Percentage of sleep efficiency was calculated by dividing the amount of time sleeping by the amount of time spent in bed. Sleep efficiency ranges from 0 to 100 percent, with higher scores indicating better outcomes.
Time Frame: Baseline to post-intervention, an average of 8 weeks
Population: The number of participants analyzed is fewer than the number of participants who completed each arm of the study due to 34 participants being lost-to-follow up and not completing sleep diaries at post-intervention.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Web-based CBT-I | Treatment as Usual
Number analyzed (Participants) | 86 | 88
percentage | 8.25317 (12.65267) | .3224638 (13.1537)

3. Secondary Outcome: Change in Sleep Duration, as Determined by Daily Sleep Logs
Description: Daily sleep diaries were used to measure sleep duration. Greater sleep duration indicates a better outcome.
Time Frame: Baseline to post-intervention, an average of 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Web-based CBT-I | Treatment as Usual
Number analyzed (Participants) | 86 | 88
hours | .3426204 (1.215072) | -.0230307 (1.191647)

4. Secondary Outcome: Change in Global Sleep Quality, as Determined by Pittsburgh Sleep Quality Index Score
Description: Global sleep quality was measured using the Pittsburgh Sleep Quality Index (PSQI). Scores range from 0 to 21, with higher scores indicating worse global sleep quality.
Time Frame: Baseline to post-intervention, an average of 8 weeks
Population: The number of participants analyzed is fewer than the number of participants who completed each arm of the study due to 27 participants being lost-to-follow up and not completing the PSQI at post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based CBT-I | Treatment as Usual
Number analyzed (Participants) | 87 | 94
units on a scale | -3.172414 (2.85383) | -.1595745 (2.926715)

5. Secondary Outcome: Change in Depression Symptom Severity, as Determined by Edinburgh Postnatal Depression Scale Score
Description: Depressive symptom severity was assessed using the Edinburgh Postnatal Depression Scale (EDPS). Scores on the EPDS range from 0 to 30, with higher scores indicating greater depressive symptom severity.
Time Frame: Baseline to post-intervention, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based CBT-I | Treatment as Usual
Number analyzed (Participants) | 89 | 94
units on a scale | -2.224719 (3.85461) | -.0425532 (3.232612)

6. Secondary Outcome: Change in Insomnia Diagnosis, as Determined by Sleep Condition Indicator
Description: Insomnia caseness (i.e., whether a participant met the Diagnostic and Statistical Manual for Mental Disorders, Fifth Edition criteria for insomnia disorder) was assessed by the Sleep Condition Indicator (SCI), which is an eight-item rating scale to screen for an insomnia diagnosis. Scores range 0-32 with higher numbers indicating better sleep quality. Participants who scored below the cutoff were defined as having insomnia caseness (≤16). The mean indicates the direction and magnitude of the preponderance of changes in that direction. That is, negative values of the mean indicate that there were more changes from a baseline SCI value between 17 and 32 to a post-intervention SCI value between 1 and 16 than changes in the other direction.
Time Frame: Baseline to post-intervention, an average of 8 weeks
Population: The number of participants analyzed is fewer than the number of participants who completed each arm of the study due to 25 participants being lost-to-follow up and not completing the SCI at post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based CBT-I | Treatment as Usual
Number analyzed (Participants) | 89 | 94
units on a scale | -.5955056 (.5160845) | -.2021277 (.5201279)

ADVERSE EVENTS:
Time Frame: Through 18 weeks after randomization.
Arm/Group | Web-based CBT-I | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/103
Other Adverse Events (participants affected / at risk) | 3/105 | 3/103
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Web-based CBT-I (N=105) | Treatment as Usual (N=103)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02805998/Prot_SAP_000.pdf